CLINICAL TRIAL: NCT04965116
Title: Progestin-Only Pill Use and Breastfeeding Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sarah Averbach, MD MAS, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 210357
Record Dates: First submitted 2021-06-26; First posted 2021-07-16 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Contraception; Breastfeeding
Keywords: Minipill; Progestin-only Pill; Postpartum; Slynd; Camila; Micronor; Infant growth; Breastmilk; Drospirenone; Norethindrone
MeSH Terms: conditions — Breast Feeding | interventions — Norethindrone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Early Initiation d-POPs (Experimental): Initiation of d-POPs 120-160 hours after delivery. Dosing is 4mg daily for 24 days followed by 4 daily inactive tablets for 2 months.
  Interventions: Drug: Progestin Only Contraceptive Pills
- Early Initiation n-POPs (Experimental): Initiation of n-POPs 120-160 hours after delivery. Dosing is 0.35mg daily for 28 days for 2 months.
  Interventions: Drug: Progestin Only Contraceptive Pills
- Interval Initiation of d-POPs (Placebo Comparator): Placebo starting 120-160 hours after delivery, continuing for 28 days. Followed by 24 days of 4mg daily of d-POPs and 4 daily inactive tablets.
  Interventions: Drug: Progestin Only Contraceptive Pills

INTERVENTIONS:
Drug: Progestin Only Contraceptive Pills — Daily pill (placebo or active tablet)
  Other Names: Slynd; Camila; Micronor; Errin

SUMMARY:
This study will assess the impact of early initiation (less than one week postpartum) and delayed initiation (4 weeks postpartum) of two types of progestin-only contraceptive pills (POPs) on maternal, breastmilk, and infant outcomes.

DETAILED DESCRIPTION:
This is a placebo-controlled randomized controlled trial enrolling dyads of birthing people and their newborn infants. We will explore if the type and timing of initiation of pills is acceptable to the user with minimal side effects, impacts the supply or composition of breastmilk, and/or affects infant growth.

Birthing people will be randomly assigned to 1 of 3 groups and will be blinded to group assignment:

1. immediate initiation of drospirenone-containing progestin-only pills (d-POPs),
2. immediate initiation of norethindrone-containing progestin-only pills (n-POPs)
3. immediate initiation of a placebo pill for one month followed by d-POPs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Desires to use POPs for 3 months
* Speak English or Spanish
* Had a vaginal or cesarean delivery of a singleton full term (≥37 weeks) infant less than 168 hours prior
* Intends to breastfeed exclusively for 6 months

Exclusion Criteria:

* Desire another pregnancy in less than 6 months
* Do not intend to exclusively breastfeed
* Do not have access to a telephone
* Have any medical contraindication to POPs
* Have any contraindication to breastfeeding, including maternal illegal drug use, history of augmentation or reduction, infant with major congenital anomaly
* Cognitively impaired
* Currently incarcerated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Averbach, MD, MAS, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Numbers represent dyads of the birthing person and infant.
Period: Overall Study
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs
Started | 10 (Dyads: birthing person and infant) | 10 (Dyads: birthing person and infant) | 10 (Dyads: birthing person and infant)
Completed | 10 (Dyads: birthing person and infant) | 10 (Dyads: birthing person and infant) | 10 (Dyads: birthing person and infant)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There are 30 total dyads enrolled, 30 birthing people and their respective 30 newborn infants. The unit of the dyad is specified for each characteristic and was either self-reported by the birthing person or collected via chart review for the infant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Birthing person
  years | 31.6 (5.6) | 31.2 (5.5) | 28.4 (3.6) | 30.4 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of the birthing person
  Participants
    Female | 10 | 10 | 10 | 30
    Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of the birthing person
  Participants
    Hispanic or Latino | 4 | 3 | 5 | 12
    Not Hispanic or Latino | 6 | 7 | 5 | 18
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of the birthing person
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 2 | 3 | 2 | 7
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 1 | 1 | 0 | 2
    White | 3 | 4 | 6 | 13
    More than one race | 1 | 1 | 0 | 2
    Unknown or Not Reported | 3 | 1 | 2 | 6
Region of Enrollment [Number; unit: birthing person/infant dyad] — Birthing person/infant dyads enrolled in the United States.
  birthing person/infant dyad
    United States | 10 | 10 | 10 | 30
Prior delivery [Count of Participants; unit: Participants] — Birthing people who have had a prior delivery.
  Participants | 2 | 3 | 4 | 9
Highest education level achieved [Count of Participants; unit: Participants] — Highest education level achieved by birthing person.
  Participants
    High school or less | 1 | 1 | 1 | 3
    Post-high school, technical school | 0 | 1 | 0 | 1
    Some college | 2 | 0 | 3 | 5
    Undergraduate degree | 5 | 6 | 2 | 13
    Some graduate degree | 0 | 0 | 1 | 1
    Completed graduate degree | 2 | 2 | 3 | 7
Using donor milk to supplement feeding in hospital [Count of Participants; unit: Participants] — Number of birthing people using donor milk to feed their infant.
  Participants | 4 | 1 | 4 | 9
Infant sex at birth [Number; unit: Infants of the dyad] — Number of infants by sex.
  Infants of the dyad
    Female | 6 | 6 | 3 | 15
    Male | 4 | 4 | 7 | 15
Infant birth length [Mean (Standard Deviation); unit: Centimeters] — Infant birth length in centimeters.
  Centimeters | 51.2 (2.1) | 51.6 (2.7) | 50.4 (2.2) | 51.06 (2.3)
Infant birth weight [Mean (Standard Deviation); unit: Grams] — Infant birth weight in grams.
  Grams | 3432 (546) | 3433 (354) | 3502 (484) | 3456 (453)
Infant birth head circumference [Mean (Standard Deviation); unit: Centimeters] — Infant head circumference in centimeters at birth.
  Centimeters | 34.3 (1.7) | 34.9 (1.5) | 35.0 (0.7) | 34.74 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Exclusive Lactation Among Birthing People at 8 Weeks Postpartum.
Description: Lactation status will be assessed at 8 weeks postpartum through an email self-reported survey.
Time Frame: 8 weeks postpartum
Population: Lactation status was reported by 22 birthing people at 8 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs
Number analyzed (Participants) | 7 | 9 | 6
Participants | 7 | 7 | 6

2. Secondary Outcome: Proportion of Birthing People Using Progestin-only Pills at 8 Weeks Postpartum
Description: Type of contraception being used at 8 weeks postpartum will be assessed through an email self-reported survey.
Time Frame: 8 weeks postpartum
Population: Progestin-only pill use was reported by 22 birthing people at 8 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs
Number analyzed (Participants) | 7 | 9 | 6
Participants | 7 | 8 | 4

3. Secondary Outcome: Vaginal Bleeding
Description: Number of days of any bleeding and spotting among birthing people in last week will be collected via self-reported email survey.
Time Frame: 8 weeks postpartum
Population: Vaginal bleeding was reported by 22 birthing people at 8 weeks.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs
Number analyzed (Participants) | 7 | 9 | 6
days | 0.1 (0.4) | 2.7 (3.1) | 0.2 (0.4)

4. Secondary Outcome: Satisfaction With Assigned POP
Description: Overall satisfaction and if birthing people would recommend the POP they were assigned to use to a friend will be ascertained from an email self-report survey. Counts are the number of birthing people who responded "yes".
Time Frame: 8 weeks postpartum
Population: Satisfaction with assigned POP was reported by 22 birthing people at 8 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs
Number analyzed (Participants) | 7 | 9 | 6
Participants | 6 | 8 | 5

5. Secondary Outcome: Protein Content of Human Milk
Description: Mid-feeding milk samples will be pumped by birthing people and analyzed.
Time Frame: 4 weeks postpartum
Population: 20 total milk samples were collected.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs
Number analyzed (Participants) | 7 | 6 | 7
ng/dL | 1.49 (0.18) | 1.46 (0.29) | 1.26 (0.28)

6. Secondary Outcome: Carbohydrate Content of Human Milk
Description: Mid-feeding milk samples will be pumped by birthing people and analyzed.
Time Frame: 4 weeks postpartum
Population: 20 total milk samples collected.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs
Number analyzed (Participants) | 7 | 6 | 7
ng/dL | 9.11 (0.61) | 8.75 (0.40) | 9.25 (1.02)

7. Secondary Outcome: Fat Content of Human Milk
Description: Mid-feeding milk samples will be pumped by birthing people and analyzed.
Time Frame: 4 weeks postpartum
Population: 20 total milk samples collected
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs
Number analyzed (Participants) | 7 | 6 | 7
ng/dL | 3.79 (0.71) | 3.53 (1.14) | 3.24 (0.61)

8. Secondary Outcome: Perception of Milk Supply
Description: Self-reported perception of adequacy of milk supply will be collected with the 20-item Hill and Humenick Lactation Scale among birthing people. Minimum scale score is 20 and maximum is 140, with higher scores representing a more positive perception of breastfeeding.
Time Frame: 8 weeks postpartum
Population: Perception of milk supply was reported by 22 birthing people at 8 weeks.
Measure: Mean (Standard Deviation); unit: Mean scale score
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs
Number analyzed (Participants) | 7 | 9 | 6
Mean scale score | 95.1 (8.0) | 96.5 (7.9) | 92.5 (6.7)

9. Secondary Outcome: Change in Infant Weight
Description: Infant weight in grams will be compared over 4 weeks.
Time Frame: Baseline and 4 weeks after delivery
Population: 20 infants weighed.
Measure: Mean (Standard Deviation); unit: Percent difference
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs
Number analyzed (Participants) | 7 | 6 | 7
Percent difference | 20.9 (13.1) | 28.4 (9.0) | 30.8 (18.7)

10. Secondary Outcome: Change in Infant Height
Description: Infant length as measured on a marked board to the nearest millimeter will be compared over 4 weeks.
Time Frame: Baseline and 4 weeks after delivery
Population: 20 infants measured.
Measure: Mean (Standard Deviation); unit: Percent difference
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs
Number analyzed (Participants) | 7 | 6 | 7
Percent difference | 7.2 (2.6) | 3.6 (4.0) | 6.8 (6.1)

11. Secondary Outcome: Change in Infant Head Circumference
Description: The maximum diameter through the infant's glabella and occiput is found and measured with a tape measure and recorded to the nearest millimeter and compared over 4 weeks.
Time Frame: Baseline and 4 weeks after delivery
Population: 20 infants measured.
Measure: Mean (Standard Deviation); unit: Percent difference
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs
Number analyzed (Participants) | 7 | 6 | 7
Percent difference | 8.4 (5.0) | 7.3 (3.8) | 7.4 (3.5)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: In this section, participants are considered individually rather than in dyads. This number equals 30 birthing people and 30 infants, making the total sample reported 60.
Arm/Group | Early Initiation d-POPs | Early Initiation n-POPs | Interval Initiation of d-POPs
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT04965116/Prot_SAP_000.pdf